CLINICAL TRIAL: NCT05049161
Title: A Long-term Extension of Study GNC-401 With Temelimab in Patients With Relapsing Forms of Multiple Sclerosis (RMS) Under Treatment With Rituximab
Brief Title: A Long-term Extension of Study GNC-401
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug product unavailability
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-402; 2021-001973-21 (EudraCT Number)
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Forms of Multiple Sclerosis; GNbAC1; Human Endogenous Retrovirus Type W; HERV-W; Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Temelimab 18 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: Temelimab 18 mg/kg
- Temelimab 36 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: Temelimab 36mg/kg
- Temelimab 54 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: Temelimab 54 mg/kg

INTERVENTIONS:
Drug: Temelimab 18 mg/kg — temelimab 18 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total)
  Arms: Temelimab 18 mg/kg
Drug: Temelimab 36mg/kg — temelimab 36 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total)
  Arms: Temelimab 36 mg/kg
Drug: Temelimab 54 mg/kg — temelimab 54 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total)
  Arms: Temelimab 54 mg/kg

SUMMARY:
This Phase II study is a monocenter, long-term extension study of study GNC-401 and will start after individual completion of Week 48 of the GNC-401 study. At entry, all patients will receive active treatment with temelimab. The patients of the placebo group in study GNC-401 will be re-randomized to temelimab 18 mg/kg, 36 mg/kg or 54 mg/kg (1:1:1), while the patients who received temelimab in study GNC-401 will continue with the same dose in study GNC-402. Following final analysis of the results of the GNC-401 study, the Sponsor may switch all patients to an optimal dose of temelimab based on safety and efficacy demonstrated in the GNC-401 study.

ELIGIBILITY:
Main Inclusion Criteria:

1. The patient has given written informed consent to participate in the study;
2. Current diagnosis of RMS, based on the McDonald 2017 criteria ;
3. Patients must have completed study GNC-401. Completion is defined as having performed the Week 48 assessments of study GNC 401;
4. Have no clinical (relapses) or MRI signs (≥2 new T2 lesions of >10 mm diameter) of acute MS disease activity, based on the Week 48 MRI of study GNC 401, or, if yes, been retreated prior to study entry with rituximab;
5. Have a B cell count ≤0.05 x 109 CD19 cells/L (assessed at the end of study GNC 401, or before inclusion in this study GNC 402 (available result from routine clinical practice); if not retreated with rituximab before entering study GNC-402, monthly B-cell count will be executed and retreatment will be considered by the treating physician when B-cells are >0.05 x 109 CD19 cells/L);

Main exclusion criteria

1. The emergence of any disease diagnosis during the course of study GNC-401 that is not due to MS and could better explain the patient's neurological signs and symptoms;
2. Body weight ≤40 kg;
3. Contraindication to continue rituximab therapy;
4. Has received rituximab less than 12 days prior to study entry;
5. Use of any of the following medications since Week 48 of the GNC 401 study:

   1. Interferon (IFN) β, glatiramer acetate, IV immunoglobulin (IVIG), dimethyl fumarate or teriflunomide;
   2. Natalizumab, mitoxantrone, cladribine, alemtuzumab, cyclophosphamide, systemic cytotoxic therapy, total lymphoid irradiation, and/or bone marrow transplantation;
   3. Highly potent immune modulating therapy, such as: ocrelizumab, ofatumumab, fingolimod, siponimod, ozanimod or anti-cytokine therapy, plasmapheresis or azathioprine;
   4. Any experimental drugs for the treatment of MS;
6. Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater lymphopenia (based on Week 48 of study GNC 401);
7. Any major medical or psychiatric disorder that would affect the capacity of the patient to fulfill the requirements of the study, including:

   1. Diagnosis or history of schizophrenia;
   2. Current diagnosis of moderate to severe bipolar disorder, major depressive disorder, major depressive episode, history of suicide attempt, or current suicidal ideation;
   3. Current or past (within the last 2 years) alcohol or drug abuse;
8. History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (New York Heart Association [NYHA] class 3 or 4);
9. Known inability to undergo an MRI scan;
10. Contraindications to the use of 5% glucose solution for infusion;
11. Inability to follow study instructions, or complete study assessments, as defined by the protocol;
12. Any history of cancer with the exceptions of basal cell carcinoma and/or carcinoma in situ of the cervix, and only if successfully treated by complete surgical resection, with documented clean margins and any medically unstable condition as determined by the Investigator;
13. Pregnant or breastfeeding women;
14. Abnormal liver function tests: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 times upper limit of normal range (ULN), or conjugated bilirubin >2 times ULN, or alkaline phosphatase (AP) or gamma-glutamyl transferase (GGT) >3 times ULN;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
safety and tolerability:adverse event | 48 weeks
  Number of Patients With Treatment-Related Adverse Events

SECONDARY OUTCOMES:
Neuroimaging | 48 weeks
  Change in Brain parenchymal volume fraction at Week 48 compared to Baseline
Neuroimaging | 48 weeks
  change in magnetization transfer Saturation (MTSat) in periventricular NAWM at at Week 48 compared to Baseline
Neuroimaging | 48 weeks
  Change in thalamic volume fraction at Week 48 compared to Baseline
Neuroimaging | 48 weeks
  Change in magnetization Transfer Saturation (MTSat) in cortex at Week 48 compared to Baseline
Neuroimaging | 48 weeks
  Change in T1 and T2 lesion volume at Week 48 compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Leppert, MD, Study Director — GeNeuro Innovation SAS
Locations (1):
- Center for Neurology, Academic Specialist Center, Stockholm, Sweden